CLINICAL TRIAL: NCT03565393
Title: Tolerability and Acceptability of Fibersol-2 (Resistant Maltodextrin) in Healthy and Diarrheal Children Followed by a Randomized Clinical Trial to Evaluate the Efficacy of Fibersol-2 in Diarrheal Children 1-3 Years Old
Brief Title: Tolerability and Acceptability of Fibersol-2 in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PR-16091
Record Dates: First submitted 2018-03-19; First posted 2018-06-21 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2018-03

CONDITIONS: Diarrhea
Keywords: Tolerability; Acceptability; Fibersol-2; Children
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: A placebo-controlled, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A placebo-controlled, randomized; double-blind 2 arm trial to assess the efficacy of fibersol-2 in children with acute watery diarrhea.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibersol-2 (Placebo Comparator): Receive Fibersol-2 twice daily
  Interventions: Combination Product: Fibersol-2
- Placebo (Placebo Comparator): Receive placebo twice daily
  Interventions: Combination Product: Fibersol-2

INTERVENTIONS:
Combination Product: Fibersol-2 — A placebo-controlled, randomized; double-blind 2 arm trial

SUMMARY:
Dietary fiber, a non-digestible carbohydrate, used in decades for the beneficial effect on health with physiological importance because such compounds have low energy values. These indigestible carbohydrates generally reach the large intestine undigested and unabsorbed, they are often used in many functional and/or low-calorie food and beverages. Researchers have stated that dietary fiber especially digestive-resistant maltodextrin has innumerable beneficial effects on human health, such as improving intestinal regularity by increasing fecal bulk, stimulating peristalsis and shortening gastrointestinal transit time. Resistant maltodextrin (Fibersol-2) is a low viscosity, water-soluble, indigestible dextrin produced by the treatment of corn starch with acid, enzymes, and heat. Dietary fiber, a non-digestible carbohydrate, has been used in decades for the beneficial effect of health with physiological importance. In developing countries most of the diarrhea episodes occur during the first two years of life and till date antibiotics have been found to have no role in over seventy five percent of young childhood diarrhea. Toddler's diarrhea which affects children aged 6 to 60 months is known as chronic nonspecific diarrhea of childhood. The stool is frequently watery or loose and may have food particles in it. Despite the diarrhea, the child continues to grow and gain weight, remains active and has a normal appetite. The beneficial effects of resistant maltodextrin are well known in developed countries; however, data are lacking in developing countries. It has become imperative to know its safety, tolerability and acceptability in small children with or without diarrhea in developing countries such as in Bangladesh.

DETAILED DESCRIPTION:
To conduct an exploratory study to understand the digestive tolerability of resistant maltodextrin (Fibersol-2) in young healthy and diarrhea children aged 1-3 years for 30 children at home and 30 children at hospital in phase 1. Additionally, propose to conduct a placebo-controlled, randomized, double blind clinical trial to examine whether Fibersol-2 with water can reduce the duration of diarrhea and stool output in children of 1-3 years old in the tertiary level hospital. If the child vomits out within 10 minutes of oral intake, we will give him again similar amount of fibersol-2 for consumption after an hour of rejection; if the child vomits again within 10 minutes of next intake, we will stop giving him fibersol-2 anymore. Also assess the digestive tolerability of the study children. In addition to gathering information from hospital, field research staff will visit the households of study children to collect information about their health status by administering field tested questionnaire.

Study staff members will follow-up the study participants round the clock (24 hrs) during their hospital stay. To ensure the patient care they maintain a roster duty with staff members consisting 2 Project Research Physicians, 4 Study Nurse, 2 Field Research Assistants and 4 Field Organizer. Project physician will be responsible for consenting as well as all clinical assessment including the assessment of the diarrheal patients and provide treatment, besides these they will be given treatment for other illness if needed, our study nurses are responsible for recording vital signs and will feed the Fibersol-2 to the study participants in front of their legal guardians at hospital and community level with appropriate dose and time. They will also be closely monitoring the participants after oral intake of fibersol-2; if any adverse event is observed they will call the study physician immediately. Field Research assistant and Field Organizer will be screening the community control as well as will record other socio-demographic information and anthropometry as required. Also assist the study nurse in monitoring the study participants at household level.

Eligibility criteria for the clinical efficacy trial

Inclusion criteria:

(i) Children with acute watery diarrhea, 3 or more watery stool in any 24-hour period of <7 days duration with none or some dehydration (ii) Aged between 1-3 years, and (iii) Received written consent from parents

Exclusion criteria:

(i) Children with bloody diarrhea, severe diseases (severe sepsis, meningitis, severe pneumonia with respiratory distress requiring intensive care and ancillary support such as oxygen inhalation, orophryngeal suction etc., (ii) Child in a situation and could interfere with the optimal participation to the study or constitute a particular risk of non-compliance, (iii) Currently participating in another clinical trial, and (iv) Parents refused to give written consent.

Methods for clinical efficacy trial

A placebo-controlled, randomized; double-blind 2 arm trial to assess the efficacy of fibersol-2 in children with acute watery diarrhea. Children with acute watery diarrhea, 3 or more watery stool in any 24-hour period of <7 days duration with no dehydration.

Study group 1, 46 will receive Fibersol-2 disolved in 50 ml drinking water, twice daily (suitable dose from the tolerability and acceptability trial)

Study group 2, 46 will receive Placebo (regular maltodextrin) disolved in 50 ml drinking water twice daily (same dose as Fibersol-2)

An experienced researcher at icddr,b, not involved in the study, will prepare the randomization list using the randomization table. The name of random allocation will be indicated on a slip of paper, kept inside the sealed envelope. The sealed envelopes will be supplied to the researcher to supply the intervention package. The children with no dehydration or some dehydration will be randomized immediately after admission.

Baseline information Children fulfilling the eligibility criteria will stay in the hospital throughout the study period until discharged. Research physician will take a detailed medical history of the enrolled children to determine the duration of and type of diarrhoea and its frequency; duration and frequency of vomiting; and presence of other symptoms such as fever, feeding difficulties, and treatment received for the illness before admission; and perform a thorough physical examination including assessment of dehydration according to the guidelines used in icddr,b and also the nutritional status will be measured and recorded.

Case management Dehydration will be assessed according to the modified WHO guidelines followed in the hospital. In children with some dehydration, the fluid deficit will be corrected with ORS in an amount 10 ml/kg/hour for the first hours, then 5 ml/kg/hr until the deficit is corrected. In addition, ongoing stool losses will be replaced with ORS 5-10 ml/kg after each watery stool. For high purging children, the ORS intake will be adjusted according to the ongoing stool loss. ORS therapy will continue until diarrhoea stops. Mothers will be advised to continue breastfeeding.

Measurements Fluids intakes (IV, ORS, and water) ORS will be given to the after measuring with a calibrated cylinder and the amount intake will be recorded every 6 hours, in case of any leftover that will be deducted from previous order. Water intake will also be measured in a similar way. When needed IV fluid will be infused through a calibrated soluset, the amount infused will be recorded every 6 hours if the child requires IV fluid therapy.

Output (stool, urine and vomitus) Stool will be collected in a bucket of known weight beneath the cholera cot with a central hole and will be measured every 6 hours with an electronic scale of a precision of 1 gram. Urine will be collected by pediatric urine collector (PUC bag) and measured with a calibrated cylinder in ml. Vomitus will be collected in a pre-weighed bowl and measured with an electronic scale. The children will be offered a defined food of known calorie after measuring with an electronic scale of precision 1 g. Any leftover will be measured and subtracted from the amount offered and amount ingested will be recorded every 6 hours. Nude body weight will be measured at admission, after rehydration, and every 6 hours until recovery from diarrhoea and then at the end of every 24 hours and at discharge. Clinical evaluation will be performed every morning and evening. Resolution of diarrhea will be defined as the passage of two consecutive soft/formed stools or no stool for 24 hours. Therapeutic success will be defined as the cessation of diarrhea within 7 days of inclusion in the study treatment. Duration of diarrhea will be calculated in hours from the time of randomization to the last watery or loose stool within 7 days. Children will be considered withdrawn from the study if their parents or legal guardian withdraw consent, or the child is withdrawn from study for treatment of any complications; data (intakes and outputs) of such children up to the time of withdrawal will be included in the analysis (intent to treat analysis). Data of the children who failed to recover within seven days (study period) will also be included in the analysis for a maximum of seven days; those will be labelled as therapeutic failures and will be treated in the hospital until recovery.

Primary outcome measures will be; duration of diarrhea, proportion of patients recovered within 72 hours, and daily stool output.

Definitions Abdominal distension occurs when substances, such as air (gas) or fluid, accumulate in the abdomen causing its outward expansion beyond the normal girth of the stomach and waist. It will be evaluated by regular measurement of abdominal girth. No set parameters for abdominal distension. To measure the abdominal girth before the IP and repeat measurement daily. If there is change that is increase in diameter of girth measurement then we will define distension. Recurrent abdominal pain or discomfort at least 3days/month in the last 3 months. [28, 29]

Abdominal pain: Abdominal pain is felt in the part of the trunk below the ribs and above the pelvis. Abdominal pain comes from organs within the abdomen or organs adjacent to the abdomen. It will be measured by asking mother's perception whether the child had the history of cry, irritability which was associated with abdominal pain. [28] Rumbling: A stomach rumble, also known as a bowel sound or peristaltic sound, is a rumbling, growling or gurgling noise produced by movement of the contents of the gastro-intestinal tract as they are propelled through the small intestine by a series of muscle contractions called peristalsis. It will be measured both by taking history from the parents and by abdominal auscultation.

Bloating: Bloating is the presence of abnormal general swelling, or increased in diameter of the abdominal area. Recurrent feeling of bloating or visible distension at least 3 days/month in the last 3 months [28]. It will also be evaluated by regular measurement of abdominal girth.

Flatulence: "flatus expelled through the anus" or the "quality or state of being flatulent", which is defined in turn as "marked by or affected with gases generated in the intestine or stomach; likely to cause digestive flatulence". It will be measured by taking history from the parents.

Stool consistency: Appearance of the stool; such as formed, mucoid, or liquid. This will be measured by direct visualization by the parents as well treating physicians.

ELIGIBILITY:
Inclusion Criteria:

* Children with acute watery diarrhea, 3 or more watery stool in any 24-hour period of <7 days duration with none or some dehydration
* Aged between 1-3 years, and
* Received written consent from parents

Exclusion Criteria:

* Children with bloody diarrhea, severe diseases (severe sepsis, meningitis, severe pneumonia with respiratory distress requiring intensive care and ancillary support such as oxygen inhalation, orophryngeal suction etc.
* Child in a situation and could interfere with the optimal participation to the study or constitute a particular risk of non-compliance
* Currently participating in another clinical trial, and
* Parents refused to give written consent.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | 72 hours
  Main outcome measure is duration of diarrhea
Stool consistency. | 24 hrs
  Stool consistency measured by regular observation

CONTACTS AND LOCATIONS:
Overall Officials: Mohammod Jo Chisti, MMed PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Kumudini Medical College and hospital, Mirzapur, Tangail, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hillemeier C. An overview of the effects of dietary fiber on gastrointestinal transit. Pediatrics. 1995 Nov;96(5 Pt 2):997-9. PMID 7494680
- [Result] Kishimoto Y, Kanahori S, Sakano K, Ebihara S. The maximum single dose of resistant maltodextrin that does not cause diarrhea in humans. J Nutr Sci Vitaminol (Tokyo). 2013;59(4):352-7. doi: 10.3177/jnsv.59.352. PMID 24064737
- [Result] Livesey G. Tolerance of low-digestible carbohydrates: a general view. Br J Nutr. 2001 Mar;85 Suppl 1:S7-16. doi: 10.1079/bjn2000257. PMID 11321031
- [Result] Bonnema AL, Kolberg LW, Thomas W, Slavin JL. Gastrointestinal tolerance of chicory inulin products. J Am Diet Assoc. 2010 Jun;110(6):865-8. doi: 10.1016/j.jada.2010.03.025. PMID 20497775
- [Result] Castillejo G, Bullo M, Anguera A, Escribano J, Salas-Salvado J. A controlled, randomized, double-blind trial to evaluate the effect of a supplement of cocoa husk that is rich in dietary fiber on colonic transit in constipated pediatric patients. Pediatrics. 2006 Sep;118(3):e641-8. doi: 10.1542/peds.2006-0090. PMID 16950955
- [Result] King DE, Mainous AG 3rd, Lambourne CA. Trends in dietary fiber intake in the United States, 1999-2008. J Acad Nutr Diet. 2012 May;112(5):642-8. doi: 10.1016/j.jand.2012.01.019. Epub 2012 Apr 25. PMID 22709768
- [Result] McGill CR, Fulgoni VL 3rd, Devareddy L. Ten-year trends in fiber and whole grain intakes and food sources for the United States population: National Health and Nutrition Examination Survey 2001-2010. Nutrients. 2015 Feb 9;7(2):1119-30. doi: 10.3390/nu7021119. PMID 25671414
- [Result] Fastinger ND, Karr-Lilienthal LK, Spears JK, Swanson KS, Zinn KE, Nava GM, Ohkuma K, Kanahori S, Gordon DT, Fahey GC Jr. A novel resistant maltodextrin alters gastrointestinal tolerance factors, fecal characteristics, and fecal microbiota in healthy adult humans. J Am Coll Nutr. 2008 Apr;27(2):356-66. doi: 10.1080/07315724.2008.10719712. PMID 18689571
- [Result] Ye Z, Arumugam V, Haugabrooks E, Williamson P, Hendrich S. Soluble dietary fiber (Fibersol-2) decreased hunger and increased satiety hormones in humans when ingested with a meal. Nutr Res. 2015 May;35(5):393-400. doi: 10.1016/j.nutres.2015.03.004. Epub 2015 Mar 18. PMID 25823991
- [Result] Guimaraes EV, Goulart EM, Penna FJ. Dietary fiber intake, stool frequency and colonic transit time in chronic functional constipation in children. Braz J Med Biol Res. 2001 Sep;34(9):1147-53. doi: 10.1590/s0100-879x2001000900007. PMID 11514838
- [Result] Gibson GR, Roberfroid MB. Dietary modulation of the human colonic microbiota: introducing the concept of prebiotics. J Nutr. 1995 Jun;125(6):1401-12. doi: 10.1093/jn/125.6.1401. PMID 7782892
- [Derived] Shahid ASMSB, Ahmed S, Dash S, Kishimoto Y, Kanahori S, Ahmed T, Faruque ASG, Chisti MJ. Is Fibersol-2 efficacious in reducing duration of watery diarrhea and stool output in children 1-3 years old? A randomized, parallel, double-blinded, placebo-controlled, two arm clinical trial. PLoS One. 2023 Jan 27;18(1):e0280934. doi: 10.1371/journal.pone.0280934. eCollection 2023. PMID 36706123
- [Derived] Shahid ASMSB, Ahmed S, Renesa TT, Onni AT, Dash S, Kishimoto Y, Kanahori S, Ahmed T, Faruque ASG, Chisti MJ. Digestive tolerability and acceptability of Fibersol-2 in healthy and diarrheal children 1-3 years old at a rural facility, Bangladesh: Results from a four arm exploratory study. PLoS One. 2022 Sep 19;17(9):e0274302. doi: 10.1371/journal.pone.0274302. eCollection 2022. PMID 36121843